CLINICAL TRIAL: NCT06517199
Title: Randomized Placebo-controlled Study of Olanzapine for Cancer Related Anorexia-cachexia Syndrome
Brief Title: Olanzapine for Cancer Related Anorexia-cachexia Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 980/2566(IRB1)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Anorexia; Cachexia
Keywords: cancer anorexia; olanzapine
MeSH Terms: conditions — Anorexia; Cachexia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): placebo 1 tablet/day for 28 days
  Interventions: Drug: Placebo
- olanzapine 2.5 (Active Comparator): olanzapine 2.5 mg/day for 28 days
  Interventions: Drug: Olanzapine 2.5 MG
- olanzapine 5 (Active Comparator): olanzapine 5 mg/day for 28 days
  Interventions: Drug: Olanzapine 5 MG

INTERVENTIONS:
Drug: Olanzapine 2.5 MG — olanzapine 2.5 mg/day for 28 days
  Other Names: OLN2.5
  Arms: olanzapine 2.5
Drug: Olanzapine 5 MG — olanzapine 5 mg/day for 28 days
  Other Names: OLN5
  Arms: olanzapine 5
Drug: Placebo — placebo 1 tab/day for 28 days
  Other Names: PLC
  Arms: placebo

SUMMARY:
Cancer anorexia-cachexia syndrome is one of the common conditions in cancer patients. Olanzapine has been demonstrated to reduce chemotherapy-induced anorexia. However, there is scarce information regarding olanzapine as a treatment of cancer anorexia among patients who does not receive chemotherapy. Therefore, this randomized controlled trial aims to evaluate the efficacy of olanzapine to lessen cancer cachexia-anorexia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* pathologically or cytologically metastatic or locally advanced cancer
* anorexia and >=5% weight loss during the past 6 months or anorexia with numerical scale of anorexia >=5
* ECOG performance status 0-3
* able to complete questionaire and able to swallow pills

Exclusion Criteria:

* receiving chemotherapy or anti-cancer systemic therapy
* life expectancy longer than 1 month
* received radiotherapy at head/neck or thoracic or upper abdomen in the past 2 weeks
* surgery within 4 weeks
* pregnancy
* serum bilirubin > 2 mg/dl or serum Cr > 2 mg/dl
* current use of olanzapine or other antipsychotic drug
* known cardiac arrhythmia, uncontrolled brain metastasis, history of seizure or acute coronary event in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
no greater than 5% weight loss in olanzapine 2.5 mg versus placebo | 4 weeks
  proportion of patients with olanzapine 2.5 mg without greater or equal to 5% weight loss compared to placebo

SECONDARY OUTCOMES:
no greater than 5% weight loss in olanzapine 5 mg versus placebo | 4 weeks
  proportion of patients with olanzapine 5 mg without greater or equal to 5% weight loss compared to placebo
numerical scale of anorexia | 4 weeks
  proportion of patients with decreased numerical scale of anorexia
body weight | week 2 and 4
  body weight change from baseline
adverse effects | week 1, 2, 3, 4
  adverse effects

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Division of medical oncology, department of medicine Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No
not yet decided

REFERENCES:
- [Background] Navari RM, Brenner MC. Treatment of cancer-related anorexia with olanzapine and megestrol acetate: a randomized trial. Support Care Cancer. 2010 Aug;18(8):951-6. doi: 10.1007/s00520-009-0739-7. Epub 2009 Sep 11. PMID 19756773
- [Background] Sandhya L, Devi Sreenivasan N, Goenka L, Dubashi B, Kayal S, Solaiappan M, Govindarajalou R, Kt H, Ganesan P. Randomized Double-Blind Placebo-Controlled Study of Olanzapine for Chemotherapy-Related Anorexia in Patients With Locally Advanced or Metastatic Gastric, Hepatopancreaticobiliary, and Lung Cancer. J Clin Oncol. 2023 May 10;41(14):2617-2627. doi: 10.1200/JCO.22.01997. Epub 2023 Mar 28. PMID 36977285
- [Background] Arends J, Strasser F, Gonella S, Solheim TS, Madeddu C, Ravasco P, Buonaccorso L, de van der Schueren MAE, Baldwin C, Chasen M, Ripamonti CI; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Cancer cachexia in adult patients: ESMO Clinical Practice Guidelines☆. ESMO Open. 2021 Jun;6(3):100092. doi: 10.1016/j.esmoop.2021.100092. PMID 34144781
- [Background] Roeland EJ, Bohlke K, Baracos VE, Bruera E, Del Fabbro E, Dixon S, Fallon M, Herrstedt J, Lau H, Platek M, Rugo HS, Schnipper HH, Smith TJ, Tan W, Loprinzi CL. Management of Cancer Cachexia: ASCO Guideline. J Clin Oncol. 2020 Jul 20;38(21):2438-2453. doi: 10.1200/JCO.20.00611. Epub 2020 May 20. PMID 32432946